CLINICAL TRIAL: NCT04667520
Title: Testing a Lifestyle Physical Activity Intervention for Women With Depression in Alcohol Treatment
Acronym: HEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202006-001; R01AA028186 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-12-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder; Depression
MeSH Terms: conditions — Alcoholism; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPA+Fitbit (Experimental): Participants in this group receive a Lifestyle Physical Activity intervention and are provided with a Fitbit to collect activity data
  Interventions: Behavioral: Lifestyle Physical Activity (LPA)
- Fitbit Only (Active Comparator): Participants in this group are provided with a Fitbit to collect activity data
  Interventions: Behavioral: Fitbit Only

INTERVENTIONS:
Behavioral: Lifestyle Physical Activity (LPA) — This intervention has 3 components: (1) an orientation session to LPA and using the Fitbit; (2) Six telephone physical activity counseling sessions; and (3) monitoring activity with the Fitbit, which is provided to them during their study participation.
  Arms: LPA+Fitbit
Behavioral: Fitbit Only — Participants are provided with a Fitbit during their study participation.
  Arms: Fitbit Only

SUMMARY:
The primary aim of this project is to test the efficacy of a technology-supported lifestyle physical activity (LPA) intervention for preventing relapse among women with depression engaged in alcohol treatment. Participants are randomized to either 1) LPA+Fitbit intervention or 2) Fitbit Only control condition. Follow-up assessments and EMA data will be collected.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is a significant and costly public health problem that affects one-third of the U.S. population in their lifetime. Women develop AUD more quickly and suffer a broader range of adverse alcohol-related health consequences than men. Physical activity (PA) interventions may play an important role as an alternate coping strategy for women with AUD and a means to decrease relapse.

The primary aim of this project is to test the efficacy of a technology-supported lifestyle physical activity (LPA) intervention for preventing relapse among women with depression engaged in alcohol treatment. A total of 214 women from the Alcohol and Drug Partial Hospitalization Program (ADP) at Butler Hospital with AUD and depression will be recruited and randomly assign them to either a: 1) LPA+Fitbit intervention or 2) Fitbit Only control condition. Follow-up assessments will occur at 6-weeks, end of treatment (EOT) at 3 months, and 6, 9 and 12 months. Participants will also complete 3, 10-day periods of ecological momentary assessment (EMA) during early recovery, at approximately weeks 1 & 2, 5 & 6, and again at weeks 11 & 12.

ELIGIBILITY:
Inclusion Criteria:

* female
* between 18 and 65 years of age
* score of 5 or above on the PHQ-9 (need to have a score of 1 on questions 1 OR 2)
* Are sedentary/low active (i.e. less than 150 minutes/week of moderate-intensity exercise for the past 3 months)
* are currently engaged in alcohol treatment
* own a smartphone - to allow for EMA software and Fitbit application

Exclusion Criteria:

* current DSM-5 diagnosis moderate/severe substance use disorder or anorexia or bulimia nervosa
* a history of psychotic disorder or current psychotic symptoms
* current suicidality or homicidality
* current mania
* marked organic impairment according to either the medical record or responses to the diagnostic assessments
* physical or medical problems that would not allow safe participation in a program of moderate intensity physical activity (i.e., not medically cleared by study physician)
* current pregnancy or intent to become pregnant during the next 12 weeks

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study enrolls females
Enrollment: 214 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent of sample that is abstinent from alcohol | 12 months
  Timeline Follow-back Interview will be used to determined whether participants drank any alcohol during the time frame assessed.

SECONDARY OUTCOMES:
Alcohol-Related Consequences | 12 months
  The Short Inventory of Problems will be used to measure the experience of alcohol-related consequences during the study period.
Depressive symptoms | 12 months
  Symptoms of depression, as measured by the Patient Health Questionnaire-9
Physical Activity levels | 12 months
  Objectively measured steps/day with a Fitbit
Alcohol Abstinence Self-Efficacy | 12 months
  Alcohol abstinence self-efficacy, as measured by Alcohol Abstinence Self-Efficacy Scale
Cardiorespiratory Fitness (estimated peak VO2) | 12 months
  Estimated VO2 max will be determined by the 6-minute Cycle Ergometer Exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Ana Abrantes, PhD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided